CLINICAL TRIAL: NCT03081221
Title: Verification of Endotracheal Tube Placement With Ultrasonography (USG) in Patients
Brief Title: Verification of Endotracheal Tube Placement With Ultrasonography (USG)
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ozlem Tolu Kendir, Fellow, Cukurova University
Other Study IDs: 60-68
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: USG

SUMMARY:
The purpose of this study is to verification of Endotracheal Tube Placement with Ultrasonography (USG).

DETAILED DESCRIPTION:
The purpose of this study is to verification of Endotracheal Tube Placement with Ultrasonography (USG). In this study, using of USG during verification will be compared with traditional method.

In traditional methods, after intubation, verification of endotracheal tube placement is done via to monitoring of thorax movement, checking of tube fogging, auscultation of lung and stomach, capnography and radiography.

In USG method, after intubation, verification of endotracheal tube placement is done via to using linear transducer. The probe will be placed transversely and longitudinally on the neck and in front of cricoid cartilage.

So, collected all data from two method will be compared.

ELIGIBILITY:
Inclusion Criteria:

* applied intubation patients

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 0-18 age children
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Detection of Tube | 1 year
  Tube shall be detected with Ultrasonography (USG)

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided